CLINICAL TRIAL: NCT01848327
Title: A Randomized Double-Blind Placebo-Controlled Study of Caprylic Triglyceride for Cognitive Impairment in Subjects With Multiple Sclerosis.
Brief Title: Caprylic Triglyceride for Treatment of Cognitive Impairments in Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Multiple Sclerosis Society (Other); Cerecin (Industry)
Responsible Party: Principal Investigator, Leticia Tornes, Assistant Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20120415; 5559072 (Other Grant/Funding Number: Fast Forward)
Record Dates: First submitted 2013-04-16; First posted 2013-05-07 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Relapsing Remitting MS; Secondary Progressive MS; Primary Progressive MS
Keywords: Cognition; Neuropsychology; Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — tricaprylin; caprylidene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Caprylic Triglyceride (Experimental): Caprylic Triglyceride (40 gram packet orally once a day for 90 days)
  Interventions: Dietary Supplement: Caprylic Triglyceride
- Placebo (Placebo Comparator): Placebo (40 gram packet orally once a day for 90 days)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Caprylic Triglyceride — Caprylic Triglyceride is a medical food that is used for the dietary management of the metabolic processes associated with mild to moderate Alzheimer's disease.
  Other Names: Axona
  Arms: Caprylic Triglyceride
Dietary Supplement: Placebo — Placebo (40 gram packet orally once a day for 90 days)
  Arms: Placebo

SUMMARY:
Background/Rationale: Cognitive problems are a common symptom in individuals with Multiple Sclerosis (MS). Treatment options are limited, and there is a pressing need for new interventions to treat MS-related cognitive impairment. Glucose (a type of sugar) is used to fuel the cells of the healthy brain. For people with neurological conditions such as MS, glucose is not converted into energy as efficiently as it would be in a healthy brain, which can lead to a decrease in cognitive function. Caprylic Triglyceride may work to bypass this problem by providing an alternative energy source that is metabolized in the liver and used by the brain.

Objective: To evaluate the therapeutic effects of 90 days of caprylic triglyceride on cognitive impairment in multiple sclerosis.

Design: Randomized, double blinded, placebo controlled trial of 158 subjects.

Outcome: Change in Total Learning (Trials 1-5) on the California Verbal Learning Test-2nd Edition-(CVLT-II) AND Change in Symbol Digit Modalities Test (SDMT) (at day 90

DETAILED DESCRIPTION:
Patients with all types of MS (Relapsing Remitting, Secondary Progressive, or Primary Progressive) are eligible to participate. Participants will undergo detailed cognitive assessment before initiating treatment and again after 90 days of treatment, to determine whether Caprylic Triglyceride demonstrates a benefit over placebo.

Dosage: 40 gram packet orally once a day Duration of Treatment: 90 days

Analyses: Interim analyses will be conducted after 72 subjects have completed the trial and objective STOP criteria for efficacy and futility have been defined in the protocol. Final analyses will be an intent-to-treat (ITT) analysis to evaluate each of the primary aims.

ELIGIBILITY:
Inclusion Criteria:

1. Institutional Review Board (IRB)-approved Informed Consent Form signed by patient
2. A diagnosis of MS as defined by the Revised McDonald criteria.
3. All subtypes of MS, relapsing and progressive, are eligible.
4. Males and females age 18 to 59 years old.
5. Complaints of difficulties with memory or other aspects of cognition.
6. Mini-Mental Status Exam (MMSE) score >=24 for determination of ability to provide informed consent.
7. 8th grade English reading proficiency as determined by Wide Range Achievement Test-4th edition-reading .
8. Females of childbearing potential must have a negative pregnancy test prior to entry into treatment phase and must simultaneously use two forms of effective contraception during the treatment and for one month or one menstrual cycle after discontinuation of the study medication.
9. All concomitant medication doses must be stable for at least 30 days prior to randomization and remain stable for the study duration.
10. An Expanded Disability Status Scale (EDSS) score of at least a 2.0 with a Functional System Score of at least a 2 in the Cerebral section due to decreased mentation.
11. Stable neurologic function with no multiple sclerosis relapses for at least 30 days prior to study entry.
12. No clinically significant abnormal findings on the physical examination, medical history, or clinical laboratory results during Screen.
13. Documented memory deficit as defined by a score at least 0.5 standard deviations (SD) below age- and gender-based normative values on the Total Learning Score of the CVLT-II OR a documented processing speed deficit as defined by a score of at least 1.0 SD below normative values on the SDMT.

Exclusion Criteria:

1. Any condition that would render the patient or the caregiver unsuitable for the study, or place them at substantial risk of adverse outcome.
2. Unwillingness/inability of the patient to fulfill the study requirements.
3. Evidence of major depression or a score on the BDI-II > or = 30 OR a score < 30 on BDI-II but with endorsed suicidal ideation.
4. Hypothyroidism
5. B12 deficiency
6. Diabetes (Type 1 or 2).
7. Positive rapid plasma reagin.
8. Fasting triglyceride level>2 times upper limit of normal value w/in 3 months of Study Visit 1.
9. History of malignancy of any organ system (other than localized squamous and basal cell carcinoma of the skin), treated or untreated, within the past 2 years.
10. Clinically significant renal disease or insufficiency.
11. Clinically significant hepatic disease or insufficiency.
12. Ethanol consumption greater than an equivalent of 2 oz/20 g/2 units of spirits per day OR 14 oz/140 g/14 units of spirits per week. One oz/10 g/1 unit of spirits = 6 oz/15 g/1 unit of wine = 12 oz/12 g/1 unit of beer.
13. History of current alcohol or substance abuse.
14. Known HIV infection.
15. History of head injury with loss of consciousness > 30 minutes.
16. History of inflammatory bowel syndrome.
17. History of severe irritable bowel disease.
18. History of severe gastroesophageal reflux disease.
19. History of diverticular disease.
20. Use of any investigational compound within 30 days prior to screening.
21. Prior or current use of medium chain triglycerides for medical purposes.
22. Known allergies to dairy products or soy.
23. Use of anticholinergic medication within 30 days prior to Study Visit 1.
24. Use of acetylcholinesterase inhibitors within 30 days prior to Study Visit 1.
25. Use of memantine within 30 days prior to Study Visit 1.
26. Use of stimulants within 30 days prior to Study Visit 1
27. Use of modafinil, amantadine, and dalfampridine within 30 days prior to Study Visit 1, unless the dose has been stable for 90 days prior to Study Visit 1
28. Use of orlistat within 30 days prior to Study Visit 1.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 124 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change in Total Learning (Trials 1-5) on the California Verbal Learning Test-2nd Edition (CVLT-II) (range from 0 to 80) | Baseline and 90 days
  measure of verbal learning and memory
Change in Symbol Digit Modalities Test (SDMT) (range from 0-110) | Baseline and 90 days
  measure of processing speed and attention
Number of participants reporting adverse events | Baseline and 90 days
  The number of participants experiencing adverse events in the active treatment and placebo group will be examined.

SECONDARY OUTCOMES:
Change in EDSS | Baseline and 90 days
  measure of disease severity
Change in Beck Depression Inventory -2nd edition (BDI-II) | Baseline and 90 days
  Self-report depression scale
Change in Multiple Sclerosis Quality of Life Inventory (MSQOL-54) | Baseline and 90 days
  Quality of life inventory
Change in Modified Fatigue Impact Scale (MFIS) | Baseline and 90 days
  Self-report Fatigue scale

CONTACTS AND LOCATIONS:
Overall Officials: Leticia Tornes, M.D., Principal Investigator — University of Miami
Locations (1):
- University of Miami Miller School of Medicine, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Via Publications